CLINICAL TRIAL: NCT07385001
Title: Phase Ib/II Trial of Atezolizumab (AK112) Combined With Albumin-Paclitaxel and Cisplatin as Neoadjuvant Therapy for Resectable, Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Prospective, Multicenter, Phase Ib/II Trial of Ivonescimab (AK112) Combined With Albumin-Paclitaxel and Cisplatin as Neoadjuvant Therapy for ESCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K202506-23
Record Dates: First submitted 2025-07-08; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Ivonescimab; Neoadjuvant
Keywords: Neoadjuvant; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1b-Cohort 1 (Experimental): Subjects will receive AK112 via intravenously (IV) Q3W
  Interventions: Drug: AK112
- Phase 1b-Cohort 2 (Experimental): Subjects will receive AK112 via intravenously (IV) Q3W
  Interventions: Drug: AK112
- Phase 2a (Experimental): Subjects will receive AK112 via intravenously (IV) Q3W+Albumin-paclitaxel 130 mg/m²,via intravenously (IV); carboplatin with an area under the curve (AUC) of 5 mg/ml/min, via intravenously (IV) Q3W, for a total of 3 cycles
  Interventions: Drug: AK112 + Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: AK112 — Cohort 1- AK112 10 mg/kg, every 3 weeks (Q3W), administered intravenously on day 1. Treatment will begin with the first patient. If the first patient does not experience any treatment-related safety issues, at least 24 hours will pass before the next 2 or 3 patients are treated.The dosing regimen and interval will remain unchanged for all patients
  Arms: Phase 1b-Cohort 1
Drug: AK112 — Cohort 2- AK112 dose of 20 mg/kg, every 3 weeks (Q3W), administered intravenously on day 1. Treatment will begin with the first patient. If the first patient does not experience any treatment-related safety issues, at least 24 hours will pass before the next 2 or 3 patients are treated.The dosing regimen and interval will remain unchanged for all patients
  Arms: Phase 1b-Cohort 2
Drug: AK112 + Neoadjuvant chemotherapy — Neoadjuvant chemotherapy:
  Albumin-paclitaxel 130 mg/m², intravenous infusion on days 1 and 8, every 3 weeks (Q3W), total of 3 cycles Carboplatin with an area under the curve (AUC) of 5 mg/ml/min, intravenous infusion on day 1, every 3 weeks (Q3W), total of 3 cycles
  AK112:
  Based on the data collected during the dose-escalation phase 1b
  Arms: Phase 2a

SUMMARY:
A Prospective, Multicenter, Phase Ib/II Trial of Ivonescimab (AK112) Combined with Albumin-Paclitaxel and Cisplatin as Neoadjuvant Therapy for Resectable, Locally Advanced Esophageal Squamous Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Written informed consent must be obtained before any study-related procedures are initiated.
* Age and Gender: Participants must be between 18 and 75 years of age, inclusive of both 18 and 75 years, and may be either male or female.
* Diagnosis and Stage: Participants must be histologically confirmed to have resectable, locally advanced esophageal squamous cell carcinoma (ESCC) with the following criteria:-T1 N1-N3 M0 or T2-T4a N0-N3 M0 (with T2 ≥ 2 cm or poorly differentiated).
* Lymph Node Status: No suspicious lymph nodes in the neck region (excluding lymph nodes in the upper thoracic esophageal area) as per neck ultrasound or enhanced CT scan; no evidence of systemic metastasis on imaging.
* R0 Resectability: The participant is expected to achieve R0 resection.
* Measurable Lesion: At least one measurable tumor lesion must be present.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected Survival: The participant is expected to have a survival duration of at least 3 months.
* Thyroid Function: Normal thyroid function is defined as a thyroid-stimulating hormone (TSH) level within the normal range. Participants with baseline TSH levels outside the normal range may still be eligible if total T3 (or free T3) and free T4 levels are within the normal range.
* Organ Function: Laboratory results must meet the following criteria:

Hematology (no blood transfusion or blood component or granulocyte colony-stimulating factor treatment within 14 days): Neutrophil count (NEU) ≥ 1.5 × 10⁹/L (1,500/mm³); Platelet count (PLT) ≥ 100 × 10⁹/L (100,000/mm³); Hemoglobin ≥ 90 g/L.

Liver: Total bilirubin (TBil) ≤ 1.5 × upper limit of normal (ULN); or for participants with TBil < 1.5 × ULN, direct bilirubin must be within the normal range; Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 × ULN.

Renal: Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance (CrCl) ≥ 60 mL/min (using the Cockcroft-Gault formula).

Coagulation: International Normalized Ratio (INR) ≤ 1.5; Prothrombin time (PT) or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.

Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 50%.

* Pregnancy Testing and Contraception: For screening-period eligible female participants of reproductive age, a serum pregnancy test must be negative. Female or male participants of reproductive capacity must be willing to use a reliable contraceptive method throughout the study period (i.e., from the date of informed consent to 90 days after the last dose of study drug), including but not limited to: abstinence, vasectomy in the male partner, sterilization in the female, effective intrauterine devices, and effective oral contraceptives.
* Compliance: The participant must be willing and able to comply with the study schedule, including visits, treatment regimen, laboratory tests, and other study requirements.

Exclusion Criteria:

* History of Other Malignancies: Participants who have had any other malignancy within 5 years prior to enrollment are excluded, except for those with localized or in situ malignancies such as basal or squamous cell carcinoma, superficial bladder cancer, cervical or breast intraepithelial neoplasia, or other conditions that are considered curable with local therapy.
* Prior Treatment with PD-1/PD-L1 Inhibitors or Other Immune-Modulating Drugs: Participants who have previously received treatment with PD-1/PD-L1 inhibitors or other drugs targeting T-cell receptors (e.g., CTLA-4, OX-40) or anti-angiogenic agents (e.g., bevacizumab, endostar) are excluded.
* Systemic Non-Specific Immune Modulation: Participants who have received systemic non-specific immune-modulating therapy (e.g., interleukins, interferons, thymopentin) within 2 weeks prior to the first dose of study drug, or who have used traditional Chinese medicine or herbal preparations with anti-tumor indications within 2 weeks prior to the first dose, are excluded.
* Active Autoimmune Disease Requiring Systemic Treatment: Participants with active autoimmune diseases requiring systemic treatment (e.g., using disease-modifying antirheumatic drugs, corticosteroids, or immunosuppressants) are excluded. Substitutive treatments (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered as systemic treatment.
* Brainstem, Meningeal, or Spinal Metastasis or Compression: Participants with brainstem, meningeal, or spinal metastasis, or with evidence of compression, are excluded.
* Significant Pleural, Pericardial, or Peritoneal Effusion: Participants with clinically significant pleural, pericardial, or peritoneal effusions requiring diuretic therapy and/or repeated drainage are excluded.
* Gastrointestinal Obstruction or Complications Within 6 Months of First Dose: Participants with a history of clinically significant gastrointestinal obstruction, perforation, intra-abdominal abscess, or fistula formation within 6 months prior to the first dose of study drug are excluded.
* Active Inflammatory Gastrointestinal Diseases: Participants with active inflammatory gastrointestinal diseases (e.g., Crohn's disease, ulcerative colitis, radiation enteritis, hemorrhagic enteritis, chronic diarrhea) are excluded.
* Tumor Encircling Major Vessels or Severe Necrosis/Hemorrhage: Participants with imaging findings showing tumor encircling major vessels, significant necrosis, or cavitation, and whose researchers determine that entry into the study would pose a bleeding risk, are excluded.
* Interstitial Lung Disease ≥ Grade 2: Participants with interstitial lung disease ≥ Grade 2 are excluded.
* Severe Cardiovascular Disease:

Uncontrolled hypertension or pulmonary hypertension; Unstable angina pectoris, myocardial infarction within 6 months prior to the first dose of study drug, coronary artery bypass grafting, or stent implantation; Chronic heart failure with NYHA functional class ≥ 2; Left ventricular ejection fraction (LVEF) < 50%;

* Severe arrhythmias requiring drug treatment (excluding atrial fibrillation or paroxysmal supraventricular tachycardia), such as QTcF > 450 msec in males or > 470 msec in females, complete left bundle branch block, or third-degree heart block; Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 4 weeks prior to the first dose of study drug.
* Severe Infection Within 4 Weeks Prior to First Dose: Participants with a history of severe infection (e.g., sepsis, bacteremia, or severe pneumonia) within 4 weeks prior to the first dose of study drug, or who have received systemic antimicrobial therapy for an active infection (excluding antiviral treatment for hepatitis B or C) within 2 weeks prior to the first dose, are excluded.
* Active Tuberculosis or Syphilis: Participants with known active tuberculosis (TB) or syphilis are excluded. Suspected TB cases must be ruled out with clinical evaluation.
* Positive HIV Antibody or Active Hepatitis B or C:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-01-28 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
DLT | 1 year
  Dose-limiting toxicity
Incidence and Severity of Adverse Events | 1 year
MTD | 1 year
  Maximum tolerated dose
RP2D | 1 year
  Recommended Phase II Dose
Major Pathologic Response(MPR) | up to 2 years
  Defined as a residual viable tumor percentage (RVT%) ≤ 10%

SECONDARY OUTCOMES:
Objective response rate (ORR) by RECIST v1.1 | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR
Event-Free Survival (EFS) | Up to 2 years
  EFS is defined as the time from randomization to the occurrence of any event, including disease progression, treatment discontinuation for any reason, or death.
Total survival time (OS) | Up to 2 years
  OS defined as the time from the first dose to death from any cause
Adverse Events (AE), Serious Adverse Events (SAE), and Immune-Related Adverse Events (irAE): Incidence and Severity | From the time of informed consent signed through 90 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospitial, Xi'an, Shannxi, China